CLINICAL TRIAL: NCT02420002
Title: Suture Care in the Pediatric Emergency Department: a Randomized Trial Comparing the Analgesic Efficacy of Hypnosis Versus MEOPA
Brief Title: Pediatric Emergency Suture Care: a Trial Comparing the Analgesic Efficacy of Hypnosis Versus MEOPA
Acronym: Hypno-Mo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2013/PF-01; 2014-002180-16 (EudraCT Number)
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Wounds, Nonpenetrating
MeSH Terms: conditions — Wounds, Nonpenetrating | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (MEOPA) (Active Comparator): Patients randomized to this arm will receive usual care, including MEOPA inhalation during local anesthetic injection and suturing.
  Intervention: Use of MEOPA during suturing Intervention: Stitch removal
  Interventions: Drug: Use of MEOPA during suturing; Procedure: Stitch removal
- Experimental arm (Hypnosis) (Experimental): Patients randomized to this arm will receive usual care as in the other arm, but before MEOPA inhalation is started, hypnosis will be tried. The local anesthetic injection and suturing will therefore take place under hypnosis (and MEOPA if necessary).
  Intervention: Use of Hypnosis during suturing Intervention: Stitch removal
  Interventions: Other: Use of Hypnosis during suturing; Procedure: Stitch removal

INTERVENTIONS:
Drug: Use of MEOPA during suturing — Patients randomized to this arm will receive usual care, including MEOPA inhalation during local anesthetic injection and suturing of a wound.
  Other Names: equimolar mixture of nitrous oxide and oxygen
  Arms: Usual care (MEOPA)
Other: Use of Hypnosis during suturing — Patients randomized to this arm will receive usual care as in the other arm, but before MEOPA inhalation is started, hypnosis will be tried. The local anesthetic injection and suturing of the wound will therefore take place under hypnosis (and MEOPA if necessary).
  Arms: Experimental arm (Hypnosis)
Procedure: Stitch removal — 6 to 15 days after the initial suturing, stitches will be removed according to usual procedures.

SUMMARY:
This is a therapeutic, randomized, single center, two parallel-arm trial comparing pain control via "MEOPA" (equimolar mixture of nitrous oxide and oxygen) in one arm versus "Hypnosis + MEOPA if needed" in the second arm.

The primary objective is to compare the two study arms in terms of efficacity for pain control according to the FLACC (Face Legs Activity Cry Consolability Observational Tool) behavioural scale.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the two study arms in terms of:

* Efficacity for pain relief during suturing according to other validated scales (a visual analog scale (VAS), the EVENDOL (Evaluation Enfant Douleur) scale);
* the duration of the procedure, the time between the start of the care process for pain (hypnosis or nitrous oxide) and the beginning of the suture;
* the amount of nitrous oxide administered;
* the conditions under which suturing takes place, in terms of (i) the general conditions of implementation, (ii) the need to use physical restraint, (iii) failure of the procedure and the need to resort to supplementary means of anesthesia, (iv) satisfaction of the operator and his/her perceived ease of operations, (v) satisfaction of the parents;
* the behavior of the patient during removal of the suture;
* the conditions under which suture removal takes place;
* complications related to the used treatments.

ELIGIBILITY:
Inclusion Criteria:

* The patient was informed about the implementation of the study, its objectives, constraints and patient rights
* The legal representative of the patient must have given free and informed consent and signed the consent
* The patient must be affiliated with or beneficiary of a health insurance plan
* The patient is available for 15 days of follow-up
* The patient is consulting in the emergency department for a wound requiring the completion of a suture and for which the operator considers that the use of nitrous oxide is necessary and possible.

Exclusion Criteria:

* The patient is participating in another interventional study
* The patient has participated in another interventional study in the last 3 months
* The patient is in an exclusion period determined by a previous study
* The patient and/or his/her parents (or legal representative) refuses to sign the consent
* It proves impossible to correctly inform the patient and / or his/her parents (or legal representative)
* The patient has a contra-indication (or an incompatible drug combination) for a treatment required in this study (MEOPA): intracranial hypertension, impaired consciousness, pneumothorax, high rate oxygen-dependence, facial trauma preventing mask application.
* The patient has a condition that makes hypnosis impossible: e.g. encephalopathy, deafness, communication disorders, does not speak French
* Suture requiring surgical exploration or an operating room, or general anesthesia or an ears-nose-throat, orthopedic or visceral surgeon (e.g. wound of the oral cavity, abdominal or thoracic penetrating wound, finger or palm wound requiring exploration by an orthopaedist)
* Fractures associated with wound
* Use of level II/III analgesics before the beginning of pre-suture care support

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-10-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Failure of pain control: yes/no | baseline (day 0)
  Failure of pain control as defined by:
  * The conversion of the procedure to MEOPA (for the hypnosis arm) or to sedation (for the MEOPA arm. Conversion is decided if the FLACC score at the end of the induction phase of hypnosis or for MEOPA is greater than 3 (1-3 are equivalent to mild discomfort).
  * Or a FLACC score> 3 during the period between anesthetic injection and the end of the suture.
The FLACC score | day 0, during anesthetic injection

SECONDARY OUTCOMES:
Pain as measured via a VAS score for children over six years of age | day 0, during anesthetic injection
  Score varying from 0.0 to 10.0
The EVENDOL score | day 0, during anesthetic injection
time lapsed between the beginning of the procedure and end of the suture | day 0
  Beginning of procedure: defined as either the beginning of MEOPA administration, or the beginning of hypnosis
  End of suture: the suture is declared as finished after cleaning the sutured zone, removal of drapes and placement of wound dressing
time lapsed between the beginning of the procedure and the beginning of the suture | day 0
  Beginning of procedure: defined as either the beginning of MEOPA administration, or the beginning of hypnosis
  Beginning of the suture: defined as the beginning of the first stitch
MEOPA use | day 0
  measured as litres/minute x minutes of administration
Qualitative scale for general suturing conditions | day 0
  classified as verg good, good, correct, or bad
Use of physical restraint? yes/no | day 0
Procedure failure: yes/non | day 0
  i..e, was it necessary to resort to complementary means in order to perform the suture?
Visual analog scale for operator satisfaction in relation to the performed procedure | day 0
Visual analog scale for operator's perception of the ease of the procedure | day 0
Visual analog scale for parental satisfaction concerning pain care and comfort during suturing | day 0
  Only one VAS per child
Visual analog scale for pain (only for children over 6) | during stitch removal (days 6 to 15)
The EVENDOL scale for pain | during stitch removal (days 6 to 15)
The FLACC scale for pain | during stitch removal (days 6 to 15)
Visual analog scale for operator's perception of the ease of stich removal | during stitch removal (days 6 to 15)
the child's behaviour during stitch removal | during stitch removal (days 6 to 15)
  classified as: calm; afraid but capable of self-control; complementary means required
The presence/absence of complications | day 0
  The presence/absence of at least one of the following complications: vomiting, nausea, agitation, imbalance problems, headache, persistant anesthesia at the end of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Fournier, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France